CLINICAL TRIAL: NCT00805259
Title: Promoting Mental Acuity in Elderly Populations Through Incentive for Technology Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: Pennsylvania Department of Health (Other Government); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Heather Schofield, Ph.D. Candidate, Harvard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMU HS08-605
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Cognitive Function
Keywords: cognitive function; elderly; technology; financial incentives; General maintenance of cognitive function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1. Atomistic (Active Comparator): payment for own work
  Interventions: Behavioral: Financial incentives
- 2. Altruistic (Active Comparator): payment for partner's work
  Interventions: Behavioral: Financial incentives
- 3. Team-based (Active Comparator): payment for relative performance of combined effort of each team
  Interventions: Behavioral: Financial incentives
- 4. Control (No Intervention): access to software but no financial incentives

INTERVENTIONS:
Behavioral: Financial incentives — Financial incentives based on use of software designed to promote cognitive function
  Arms: 1. Atomistic; 2. Altruistic; 3. Team-based

SUMMARY:
In this between-subject randomized controlled trial the investigators will test the impact of three novel structured financial incentives: atomistic, altruistic and team-based. These incentive schemes will be used to motivate one month of daily use of software designed to improve cognitive function (including memory, reaction times, attention and executive function) among the elderly. The 400 participants will be members of retirement communities in Pennsylvania. Three outcomes will be monitored and analyzed: activities completed using the software (primary), performance on the activities, and changes in cognitive functioning. This study is designed to be a pilot study. The investigators will have 90% power to find a mean daily difference of 4 activities completed in the control group versus 7 activities completed in the incentive groups assuming a standard deviation of 3.5 and an alpha of 0.017 (the bonferroni corrected significance level to account for multiple comparisons). In addition during a three month "follow-up period" all participants will have continued access to the software, however, no incentives will be provided for use. This period will be used to assess the impact of the initial incentives on long run use after financial incentives have ceased.

DETAILED DESCRIPTION:
The proposed study, a 4-arm randomized control trial, tests three novel incentive systems intended to promote the daily use of computer programs designed to improve memory and mental acuity among residents of retirement communities. Three outcome measures will be used to assess the effectiveness of the incentive programs: number of activities completed using the software (primary outcome of interest), performance on the activities, and differences between pre and post measures of mental acuity (using a standardized test of mental functions). Incentives to use the software will be offered to individuals in the experimental conditions for the first month of the 4 month study. After the initial month of incentives, all individuals will have continued access to the software, however, no incentives will be provided for use.

Incentives: Three incentive structures will be tested against one control group:

1. Control: Access to software programs, but no rewards for use.
2. Atomistic: Each individual is rewarded for his or her individual participation
3. Altruistic: Participants will be paired with an individual at a different retirement community and will be rewarded according to the other individual's participation
4. Combination cooperative/competitive: Individuals will be paired in teams which will compete against each other. Each team will be rewarded according to relative participation, but members within a team will receive the same amount.

Pairs will be matched on gender, age, and education, and then pairs will be randomly assigned to the different incentive conditions. Rewards in all incentive conditions will range to a maximum of $5 per day, and will be awarded differently depending on the incentive condition. Although participants will be informed of their winnings each day (to give frequent positive reinforcement), they will be paid cumulated amounts once a month (to reduce transactions costs and to ensure that actual payments are substantial). The number of activities completed using the software (up to 10 daily, or approximately 30 minutes of use) will be the basis for daily incentive payments to reward effort and avoid discouraging those who are not highly skilled. Cognitive testing will be done with the NueroTrax Mindstreams cognitive testing software.

Subjects: Roughly 400 participants will be recruited from local retirement communities which offer computing services to their residents. Subjects will be between the ages of 55 and 85 and will be required to sign informed consent forms before they are admitted to the study. Due to our focus on a population facing cognitive declines, extra care will be taken to ensure that all participants understand the information provided in the informed consent document. We will not enroll potential participants who are not able to verbalize understanding of the contents of the consent form. Participants will be trained in basic computer use and operation of the software using the Carnegie Mellon University mobile research van (see http://www.cmu.edu/news/archive/2007/June/june20_datatruck.shtml).

This pilot study will serve as the basis for a larger-scale study of financial incentives for elderly individuals to engage in mentally challenging tasks that help them improve cognitive function. In addition, this research will help us determine the relative effectiveness of different types of incentive designs that could be used in further studies of the use of financial incentives to encourage the elderly to engage in a variety of other healthy behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 85
* Resident in participating retirement community

Exclusion Criteria:

* Unstable medical conditions that would likely prevent the subject from completing the study
* Severe depression
* Inability to read or severe cognitive deficits that would preclude ability to read consent form or fill out surveys

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Daily activities completed | 4 months

SECONDARY OUTCOMES:
Performance on completed activities | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: George Loewenstein, PhD., Principal Investigator — Carngie Mellon University; Kevin Volpp, MD PhD, Principal Investigator — Univeristy of Pennsylvania and Philadelphia Bereans Administration Medical Center; Heather Schofield, Principal Investigator — Harvard University
Locations (1):
- Retirement communities near Pittsburgh Pennsylvania, Pittsburgh, Pennsylvania, United States